CLINICAL TRIAL: NCT06368336
Title: Health Related Quality of Life After Intensive Care for Sepsis, a National Cohort Study.
Status: Completed | Type: Observational
Sponsor: Uppsala University Hospital (Other)
Collaborators: Sepsisfonden (Unknown)
Responsible Party: Principal Investigator, Miklos Lipcsey, Professor, Uppsala University Hospital
Other Study IDs: 994894
Record Dates: First submitted 2024-03-25; First posted 2024-04-16 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Sepsis; Septic Shock; Sepsis, Severe
Keywords: RAND-36; ICU-treatment; Health-related Quality of Life; HRQoL; ICU-outcome; SF-36
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sepsis case: Nationwide registry of patients admitted to ICU treatment for or with sepsis, in Sweden, older than18 years of age.
- Control: Age and gender matched population controls.

SUMMARY:
The study aims to map the health-related quality of life (HRQoL) after intensive care for Sepsis with the hypothesis that it will be lower than that in the general population. The investigators also want to identify factors that are associated with low HRQoL, to see if those are available for interventions from the health care system and society to improve quality of life after treatment for sepsis in the intensive care unit (ICU).

DETAILED DESCRIPTION:
Background Sepsis is a common condition in intensive care units leading to severe illness with a high mortality. It can also lead to significant disability for the individuals after recovery.

Objective The investigators aim to study how intensive care for/with sepsis impacts the HRQoL and, if possible, identify improvable factors in the treatment and rehabilitation.

Method This is a cohort study on all ICU patients with sepsis registered in the Swedish Intensive Care registry (SIR) as well as age and gender matched population controls. The primary outcome variable HRQoL will be assessed by RAND-36. The investigators assess functional recovery by sick leave free days. SIR provides post-ICU follow-up data on RAND-36. The investigators will merge these data with data on comorbidity from the National patient register, causes of death from the National death registry, socioeconomic factors from Statistics Sweden, as well as the data on social benefits from the Swedish Social Insurance Agency.

The main analysis compares RAND-36 from sepsis patients with population controls over time. The investigators will also compare the complete sepsis cohort's burden of inability to work before and sick leave free days after sepsis with matched population controls. Additionally, the investigators will describe the complete sepsis cohort's burden of disease measured with Charlson Comorbidity Index against matched population controls.

Ethics The study has ethical permission from Swedish Ethical Review Authority, nos 2022-00445-01 and 2022-07264-02.

Eligibility All patients over 18 with sepsis or septic shock diagnosis admitted to ICU between January 1st 2008 until February 28th 2020 .

Study Population Nationwide registry of patients admitted to ICU treatment in Sweden. Intervention/Treatment No active intervention, but the study subjects have had Intensive Care for sepsis or septic shock.

Official title Health Related Quality of Life after intensive care for Sepsis, a National Cohort study.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to an ICU in Sweden that reports to the Swedish ICU register
* Admitted between January 1st 2008 until February 28th 2020
* Admitted for sepsis or septic shock and / or
* Received sepsis or septic shock diagnosis during ICU stay

Exclusion Criteria:

* Age under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Nationwide registry of patients admitted to ICU treatment in Sweden.
Sampling Method: Non-Probability Sample
Enrollment: 210484 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Health-related Quality of Life after ICU (intensive care unit) treatment with/for sepsis | Data dependent but up untill about 15 moth anticipated
  Health-related Quality of Life (HRQoL), measured with the RAND-36 test over time after ICU treatment with/for sepsis compared with population controls. The RAND-36 is a test that assess Health-Related Quality of Life were higher scores are associated with higher HRQoL.

SECONDARY OUTCOMES:
Ability to work before and after ICU (intensive care unit) treatment for Sepsis | 1 year prior ICU admittance and 2 years after ICU admittance
  The investigators will also compare the complete sepsis cohort's sick leave free days after sepsis with matched population controls. This by the Swedish Social Insurance Agency register on days with economic compensation for sick leave.
The burden of disease at ICU (intensive care unit) admittance and after ICU treatment for Sepsis | From ICU admittance and 2 years after ICU admittance
  The investigators will describe the burden of disease with Charlson Comorbidity Index according to registered diagnoses with matched population controls at ICU admittance and after ICU treatment for Sepsis. The Charlson comorbidity index is primarily used for predicted mortality rate based on comorbidity and age were higher scores predicts higher predicted mortality rate.

CONTACTS AND LOCATIONS:
Overall Officials: Miklós Lipcsey, MD, PhD, Principal Investigator — Uppsala University

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are available from the respective national registries in Sweden with restrictions as defined by the General Data Protection Regulation (GDPR), the Swedish Personal Data Act (1998:204), and the licenses with the respective national registries, and so are not publicly available. Data are however available from the respective national registries after reasonable request and adequate permissions from the Swedish ethical review authority under the restrictions outlined above.

REFERENCES:
- [Derived] Halvorsen P, Marks-Hultstrom M, Wallin E, Ahlstrom B, Lipcsey M. Health-related quality of life and functional recovery after intensive care for sepsis in a national cohort. Intensive Care Med. 2025 Jul;51(7):1282-1291. doi: 10.1007/s00134-025-07998-8. Epub 2025 Jun 23. PMID 40549021